CLINICAL TRIAL: NCT06932029
Title: Improving High Blood Pressure in Older Adults Living With Multiple Chronic Diseases - The SMBP Study
Brief Title: SMBP Study: Improving High Blood Pressure in Older Adults With Multiple Chronic Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korey Kennelty (Other)
Responsible Party: Sponsor-Investigator, Korey Kennelty, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202407611; HMC-2023C2-33427 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-03-28; First posted 2025-04-17 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMBP-pharmacist (Experimental): Self-measured blood pressure with clinical pharmacist support
  Interventions: Behavioral: SMBP with clinical pharmacist support
- SMBP-conventional (No Intervention): Self-measured blood pressure with conventional clinical support

INTERVENTIONS:
Behavioral: SMBP with clinical pharmacist support — Self-measured blood pressure with clinical pharmacist support
  Arms: SMBP-pharmacist

SUMMARY:
Nearly half of adults in the United States (47 percent, or 116 million) have hypertension, also known as high blood pressure (BP). Uncontrolled high BP can be devasting as it can lead to stroke, heart attack and kidney failure, as well as other numerous health conditions. Hypertension can be controlled; however, only one in four of adults with hypertension have their BP controlled. The chance of having high BP increases as one ages, requiring the need to examine effective hypertension strategies in older adults. The issue of hypertension management is compounded even further among older U.S. adults who live with multiple chronic diseases.

National organizations identified several effective health systems strategies for improving rates of BP control, including patient self-measured blood pressure (SMBP) monitoring. SMBP involves a patient's regular use of personal BP monitoring devices to assess and record BP across different points in time, typically at home. The evidence base for utilizing SMBP strategies in healthcare systems and practices is strong. However, there is not research regarding SMBP including how to include it into workflow in primary care clinics. Previous research has shown SMBP is beneficial, but more information is needed regarding whether SMBP is beneficial in high-risk populations (such as rural, older adults or Black, older patients).

The research team will test whether SMBP with normal clinical support vs SMBP with clinical pharmacist support improves BP in older adults living with multiple chronic conditions. The addition of a pharmacist has been shown to improve patient outcomes, though the effectiveness of SMBP with a clinical pharmacist in older adults is not known. The primary outcome will be change in systolic BP over 12 months. The secondary outcome will be self-reported treatment burden over 12 months, using a validated tool called the Multimorbidity Treatment Burden Questionnaire. The research team plans to include a subgroup of rural, older adults and Black, older adults and will not exclude older adults who have dementia.

DETAILED DESCRIPTION:
The purpose of the study is to compare the effects of self-measured blood pressure (SMBP) with conventional clinical support (SMBP-conventional) and SMBP with clinical pharmacist support (SMBP-pharmacist) on two outcomes among older adults living with multiple chronic diseases: systolic blood pressure (primary outcome), and self-reported treatment burden in selfcare (secondary outcome).

The primary outcome will be change in systolic BP after 12 months of follow-up. The primary hypothesis is that systolic BP will be significantly improved (i.e. lowered) in older adult patients living with multiple chronic diseases from primary care clinics randomized to the SMBP-pharmacist group compared to primary care clinics randomized to SMBP-conventional. The investigators further hypothesize this improvement will also occur within the two subgroups (i.e., rural, older patients and Black/African American, older patients).

STUDY DESIGN This is a multi-center, cluster-randomized, parallel-group, superiority, pragmatic trial testing two ways of addressing uncontrolled hypertension in older adults (SMBP-conventional vs SMBP-pharmacist). The investigators have designed the study to follow CONSORT 2010 guidelines for conducting randomized clinical trials. This is a pragmatic clinical trial with minimal exclusion criteria in order to facilitate the generalizability and practical application of findings. Further, the study's approach to data collection is also highly pragmatic in that primary, secondary, exploratory, and implementation outcomes as well as fidelity measures will be collected in part through clinic medical records and Medicare data. The unit of randomization is the primary care clinic with clinics stratified by healthcare system type (academic, independent, community health center). The study team chose the primary care clinic as the unit of randomization to avoid contamination within clinics that could occur with patient- or provider-level randomization.

CLINIC ELIGIBILITY AND RECRUITMENT To be eligible, clinics need to affiliate with one of the healthcare systems or practice-based research networks (PBRNs) participating in the study, provide primary care services to adults at least 65 years of age, staff providers who prescribe medications (including physicians [MDs and DOs] and advanced practice providers), and have access to patient-level electronic medical record data (for purposes of data collection and determining clinic and patient eligibility). Clinics eligible for the study will specialize in family medicine, internal medicine, or geriatrics. Clinics located in rural zip codes according to RUCA (rural-urban commuting area) categories 4-9 will be prioritized for recruitment into the study as well as clinics where at least 35% of the patients 65+ years of age are identified in healthcare system/PBRN records as Black/African American and/or identify as Black/African American in a mixed-race category.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 65 years of age
* Patient is seen at least once in clinic or healthcare system in the previous 12 months
* Patient has a six-month average (non-acute/maintenance) systolic blood pressure (SBP) >= 145 mmHg, documented in the electronic medical record in last six months
* Patient has a baseline in-clinic visit systolic blood pressure (SBP) >= 140 mmHg
* Patient plants to receive care from participating healthcare system for the next 24 months

Exclusion Criteria:

* The patient is enrolled in hospice or has an active referral to hospice care
* The patient resides in a nursing home, in skilled nursing, rehabilitation facility, or memory care
* The patient is not capable of providing informed consent
* The patient is unable to communicate in English or Spanish
* The patient is in active chemotherapy or radiation treatment for cancer
* The patient is pregnant or has plans to become pregnant
* The patient is currently participating in another study focused on blood pressure
* The patient does not have a telephone

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline and 12 months
  Change in systolic blood pressure

SECONDARY OUTCOMES:
Multimorbidity Treatment Burden Questionnaire | Baseline and 12 months
  Score range of 0-100, with 100 indicating worst outcome

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa